CLINICAL TRIAL: NCT03597477
Title: Intranasal Dexmedetomidine Combined With Oral Midazolam for Procedure Sedation in Children With Autism Spectrum Disorders During Magnetic Resonance Imaging
Brief Title: Procedure Sedation With Dexmedetomidine in Children With Autism Spectrum Disorders During Magnetic Resonance Imaging
Status: Completed | Type: Observational
Sponsor: Guangzhou Women and Children's Medical Center (Other)
Responsible Party: Principal Investigator, Ying Jun She, MD, Director, Clinical Resesearch, Department of Anesthesiology and Perioperative Medicine, Guangzhou Women and Children's Medical Center
Other Study IDs: Intranasal dexmedetomidine
Record Dates: First submitted 2018-07-10; First posted 2018-07-24 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism Spectrum Disorder; Dexmedetomidine
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Dexmedetomidine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Autism Spectrum Disorder: Patients with a diagnosis of autism spectrum disorder
  Interventions: Drug: Dexmedetomidine
- Control: Patients with no developmental diagnoses
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — participants were randomly allocated to receive sedation with oral midazolam(0.3 mg/kg) combined with 4 doses of intranasal dexmedetomidine(1.0, 1.5, 2.0, 2.5)
  Other Names: intranasal dexmedetomidine

SUMMARY:
Autism spectrum disorders (ASD) is a neurodevelopmental disorder and is characterized by functional impairment in social communication, restricted interests, and repetitive behaviors.The children with ASD has been shown different drug responses from the normal population of children. The children with ASD maybe more prone to elevate anxiety and the difficult of sedation during MRI scanning.The purpose of this investigation was to compare the effectiveness of dexmedetomidine sedation in children with and without ASD undergoing MRI scanning.

DETAILED DESCRIPTION:
The use of medications in adolescents and young adults with ASD is extremely common. However, few data address the effectiveness and harms of medications for procedural sedation in this population. It's advisable to be used as a first line medication with alpha-2 agonists for procedure sedation. The primary goal of this study was to compare the effectiveness of dexmedetomidine sedation, also determine the 50% and 95% effective doses in children with and without ASD undergoing MRI scanning.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I or II,
* Patients aged 2 years through 12 years of age scheduled for procedure sedation during MRI scanning
* Patients must have a diagnosis of Autism Spectrum Disorder (ASD) according to the DSM V (autism group) or no history of neurodevelopmental concerns (control group). Child in control group is matched to an autism spectrum disorder participant according to age, gender, and ASA level.

Exclusion Criteria:

* Known allergy or hypersensitive reaction to dexmedetomidine
* Organ dysfunction, and significant developmental delays or behavior problems
* Cardiac arrhythmia
* Known. acyanotic congenital heart disease or children after cardiac interventional procedures for follow-up examination

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children undergoing MR scanning at Guangzhou Women and Children Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 136 (Actual)
Dates: Start 2018-07-16 (Actual); Primary Completion 2020-09-17 (Actual); Study Completion 2020-09-18 (Actual)

PRIMARY OUTCOMES:
The 50% and 95% effective doses of intranasal dexmedetomidine | up to 1 hours after MRI scanning
  Children were randomly allocated to receive sedation with 1 of 4 doses (1.0, 1.5, 2.0, and 2.5 ug/kg) of dexmedetomidine. Sedation status was evaluated by a attending anesthesiologists every 5-10 min with a 6-point sedation scale, which was modified from the Modified Observer Assessment of Alertness and Sedation Scale (MOAA/S).Successful sedation was defined as an MOAA/S of between 0 and 3. Probit analysis (linear regression plot of log concentration vs percentage response) was used to estimate the 50% and 95% effective concentration values of dexmedetomidine.
  MOAA/S scale:
  0 Does not respond to a noxious stimulus
  1. Does not respond to mild prodding or shaking
  2. Responds only after mild prodding or shaking
  3. Responds only after name is called loudly or repeatedly
  4. Lethargic response to name spoken in normal tone
  5. Appears asleep, but responds readily to name spoken in normal tone
  6. Appears alert and awake, responds readily to name spoken in normal tone

SECONDARY OUTCOMES:
sedation induction time | up to 45 min after drug administration
  Successful sedation was defined as an MOAA/S of between 0 and 3, and sedation induction time was defined as the time from midazolam and dexmedetomidine administration to the onset of satisfactory sedation
Wake -up time | up to 4 hours after drug administration
  Children were classified as awake if the MOAA/S was between 4 and 6. Wake -up time was defined as the time from successful sedation until the time that the child awoke

CONTACTS AND LOCATIONS:
Overall Officials: Ying-Jun She, MD., Principal Investigator — Guangzhou Women and Children Medical Center
Locations (1):
- Guangzhou Women and Children Medical Center, Guangzhou, Guangdong, China